CLINICAL TRIAL: NCT04061018
Title: The Genetic, Protein, and Lipid Basis of Variation in Cholesterol Efflux
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anand Rohatgi, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 042016-020; 1R01HL136724-01A1 (NIH)
Record Dates: First submitted 2019-07-26; First posted 2019-08-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lipid Metabolism Disorders
Keywords: HDL; Atherosclerotic Cardiovascular Disease; Cholesterol efflux
MeSH Terms: conditions — Lipid Metabolism Disorders; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High Cholesterol Efflux: Dallas Heart Study participants who are above the sex and ethnicity specific 90th % of cholesterol efflux
- Low Cholesterol Efflux: Dallas Heart Study participants who are below the sex and ethnicity specific 10th % of cholesterol efflux

SUMMARY:
The rationale of this research is that deep phenotyping of individuals at the extremes of cholesterol efflux will identify key determinants of efflux that are potential novel therapeutic targets to prevent or reverse Atherosclerotic Cardiovascular Disease (ASCVD). The investigators propose to carry out the objective by studying participants at extreme low and high cholesterol efflux identified from the investigator's study in the population-based Dallas Heart Study by accomplishing the following aims: 1) determine the heritability of and genomic factors associated with cholesterol efflux by establishing a family pedigree of extreme low and high efflux and sequencing candidate genes involved in HDL metabolism; and 2) identify the protein and lipid signature of extreme low and high cholesterol efflux in a sex- and ethnicity-specific manner using mass spectroscopy and ELISA in FPLC-derived fractions. The investigators expect to identify genetic variants and sex- and ethnicity-specific combinations of proteins and lipids in participants with extreme low and high efflux that may lead to novel ways to modulate efflux. This proposal leverages a well-phenotyped population-based study to characterize the gene-protein-lipid signature of 1) extremes of cholesterol efflux in a sex- and ethnicity-specific manner. Successful completion of these aims will have immediate and direct impact on the use of cholesterol efflux as a clinically relevant biomarker of therapeutic benefit and are necessary for the clinical development of appropriate new targets for manipulation of the key atheroprotective function of cholesterol efflux to reduce ASCVD.

DETAILED DESCRIPTION:
The mechanisms that underlie variation in cholesterol efflux are unknown. There is a critical need to identify factors that regulate cholesterol efflux to effectively advance the clinical development of cholesterol efflux as both a risk prediction marker and as a target of therapy. The investigator's long-term goal is to determine whether modulating cholesterol efflux prevents or reverses cardiovascular disease. The overall objective of this study is to systematically create a family pedigree and biobank repository of blood and DNA from participants from the Dallas Heart Study with extreme low or high cholesterol efflux, with the specific aims of : 1) determining the heritability of and genomic factors associated with cholesterol efflux, and 2) identifying the protein and lipid signature of extreme low and high cholesterol efflux in a sex- and ethnicity-specific manner. The investigator's central hypothesis is that a combination of genetic variation in lipid transporters as well as proteins and lipids will be most strongly correlated with variation in efflux.

DHS probands and their relatives (parents, siblings, adult children, grandparents, aunts/uncles, cousins) with extreme low or high cholesterol efflux will be recruited to establish a prospective family pedigree cohort and understand the heritability of extreme cholesterol efflux. Investigators will collect the following information from all participants: demographics, health history, lifestyle measures, and medications. Blood will be collected on-site by venipuncture and plasma, serum, and cells will be stored at -80o Celsius. All efflux measurements will be completed in the investigator's laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Dallas Heart Study (DHS) Participants who are above or below the sex- and ethnicity-specific 10th and 90th% of cholesterol efflux.
* Family members of the DHS participants are also eligible

Exclusion Criteria:

* HIV
* Cancer
* Autoimmune diseases
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from the Dallas Heart Study (DHS) with extreme low or high cholesterol efflux will be recruited in this study. DHS is a multi-ethnic, population based probability sample of Dallas County designed to define the social and the biological variables contributing to ethnic differences in cardiovascular health at the community level.
  https://www.utsouthwestern.edu/edumedia/edufiles/research/center_translational_medicine/dallas_heart_study/dhs-study-overview.pdf
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Contribution of genetic factors to variability in cholesterol efflux | Anticipated completion date - November 2022
  The expected outcome is establishing the degree of heritability of the extreme low or high cholesterol efflux phenotype, specific for sex and ethnicity and the contribution of common and rare genetic variants to cholesterol efflux. This will establish for the first time to what degree inherited verses environmental factors associate with variation in cholesterol efflux.
Circulating metabolites and proteins linked to variation cholesterol efflux | Anticipated completion date - November 2022
  The investigators will measure circulating metabolites and proteins and identify the most relevant to the high/low cholesterol efflux phenotype, offering the potential to focus future studies targeting metabolic regulators of efflux.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Rohatgi, MD, Principal Investigator — UT Southwetsern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States